CLINICAL TRIAL: NCT07279480
Title: Household Communication and Health Investments for Elderly Women in Tamil Nadu
Brief Title: Communication and Health Investments for Elderly Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2505001660
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Take-up of Preventative Care; Communication About Health Information
Keywords: Elderly women; India; Household communication; Preventative health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tell elder only, without transport (Control) (No Intervention): Elder is informed about the check-up. No free arranged transportation offered.
- Tell elder only, with free transport (Experimental): Elder is informed about the check-up. We offer to arrange private transportation to and from the hospital at no cost.
  Interventions: Behavioral: Free Transport
- Tell elder and caretaker, without transport (Experimental): Both elder and the caretaker are directly informed about the check-up. No free arranged transportation offered.
  Interventions: Behavioral: Tell both
- Tell elder and caretaker, with free transport (Experimental): We offer to arrange private transportation to and from the hospital at no cost.
  Interventions: Behavioral: Tell both; Behavioral: Free Transport

INTERVENTIONS:
Behavioral: Tell both — Both elder and the caretaker are directly informed about the check-up.
  Arms: Tell elder and caretaker, with free transport; Tell elder and caretaker, without transport
Behavioral: Free Transport — We offer to arrange private transportation to and from the hospital at no cost.
  Arms: Tell elder and caretaker, with free transport; Tell elder only, with free transport

SUMMARY:
This study investigates how household communication plays a role in elderly women's take-up of health check-ups in rural Tamil Nadu, India. First, we survey elders and their caretakers to measure demand for check-ups for elders. We measure how interest in check-ups changes when we offer different versions of transportation support, to understand how much interest in check-ups are affected by the degree of caretaker involvement required. Second, we conduct a randomized evaluation of interventions to improve take-up of free health check-ups at a nearby private hospital. We will cross-randomize two interventions. The first randomizes who is informed about the check-up: either only the elder is informed or both the elder and the caretaker are informed about the check-up. The second randomizes whether free transportation is provided to and from the check-up. We will measure take-up of the check-up. We will also measure elders' willingness to mention the check-up to the caretaker.

ELIGIBILITY:
Inclusion Criteria:

* Elderly women aged 60-75

Exclusion Criteria:

* Those with severe hearing, speech, mental, or mobility impairment

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Sign-up rates for check-up. | Assessed at 3 days after the intervention
  This will be a measure of whether the elder is signed up for the check-up by the caretaker. This will be measured either when the caretaker calls to reserve a spot for the elder or when the research team follows up with the household before the check-up.

SECONDARY OUTCOMES:
Elder attendance at check-up. | 1 week after the intervention
  This is a measure of whether the elder shows up to the health check-up at the end of the week. Attendance at the health check-up will be measured by surveyors at the hospital, about 1 week after the health check-up invitations are shared with households.
Elder willingness to mention check-up to caretaker | Assessed 2 days after the intervention
  This is a measure of whether elder chooses to mention check-up to caretaker when offered. Among elders in households that are randomized into the "Tell elder only" arm, we will offer to inform the caretaker of the check-up on behalf of the elder and record whether the elder was willing to have us mention the check-up as one of our outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL SA at IFMR, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No